CLINICAL TRIAL: NCT06933979
Title: Changes in the Position of Mandibular Third Molar in Orthodontically Treated Patients With First Premolars Extraction
Brief Title: Positional Changes of Mandibular Molar After Orthodontic Treatment
Status: Active, not recruiting | Type: Observational
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, Shereen Aly El-Mahlawy, lecturer, Fayoum University
Other Study IDs: wisdom
Record Dates: First submitted 2025-03-26; First posted 2025-04-18 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Third Molar
Keywords: orthodontic treatment; premolar extraction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This retrospective study was carried out on pre and posttreatment digital standardized panoramic radiographs of 30 cases previously orthodontically treated with four first premolar extraction.

ELIGIBILITY:
Inclusion Criteria:

- class I malocclusion cases (0 < ANB < 4) with moderate crowding

Exclusion Criteria:

* Absence of all permanent teeth including mandibular third molars.

Ages: 14 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Sample size calculation estimated the minimum total required sample size (n) was found to be (27). The sample size was increased to (30) account for sample variability and to improve the robustness of statistical testing
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2025-02-23 (Actual); Primary Completion 2025-04-20 (Estimated); Study Completion 2025-04-25 (Estimated)

PRIMARY OUTCOMES:
Assessment of mandibular third molar positional variation | 2 years
  measure angles:• LA-ISL: The inward angle (towards the 2nd molar) between long axis of mandibular third molar and the inter-sigmoid line (line connecting the deepest point of the right and left sigmoid notch of the mandible).
  • LA-IMB: The inward angle between long axis of mandibular third molar and the inferior border of the mandible.

CONTACTS AND LOCATIONS:
Overall Officials: Shereen A Mahlawy, PHD, Principal Investigator — lecturer of orthodontics, faculty of dentistry, Fayoum university; clinical cT trial, Study Director — Clinical trials.gov
Locations (1):
- Fayoum University, Al Fayyum, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Zarin DA, Tse T, Williams RJ, Califf RM, Ide NC. The ClinicalTrials.gov results database--update and key issues. N Engl J Med. 2011 Mar 3;364(9):852-60. doi: 10.1056/NEJMsa1012065. PMID 21366476